CLINICAL TRIAL: NCT05701371
Title: NON-INTERVENTIONAL STUDY, MULTICENTRIC STUDY, AIMING AT CONSTITUTING A BIOLOGICAL SAMPLES COLLECTION FROM CENTENARIAN PEOPLE
Brief Title: BACTERIA ISOLATION FROM STOOLS COLLECTED FROM CENTENARIANS PEOPLE
Acronym: BISCOTE
Status: Terminated | Type: Observational
Why Stopped: Recruitment issues
Sponsor: Bioaster (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A02293-40
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Healthy Aging
Keywords: Biobank; Observational Study; Blood; Feces; Probiotics; Strain Isolation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood + Stools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Centenarian cohort
  Interventions: Other: Biological samples collection

INTERVENTIONS:
Other: Biological samples collection — blood drawing + feces collection in a dedicated device

SUMMARY:
The compositional analysis of commensal bacterial populations collected from a variety of clinical samples has been recently made possible with the availability of Next Generation Sequencing (NGS) technologies. The term 'next-generation probiotics' (NGP) is now widely used to describe these commensal species of potential health interest. However, this approach is still hampered by the fact that there are usually few or even no strains available for a number of commensal species. In this context, BIOASTER has developed a specific technological process based on flow cytometry analysis and then sorting under strictly anaerobic conditions to target and cultivate commensal species of interest.

The review of the literature shows that certain species present among centenarians have an interest in maintaining the longevity of these individuals. Numerous studies have shown that the intestinal microbiota of centenarians presents a greater diversity compared to groups of younger subjects as well as an enrichment in certain bacteria such as Akkermansia and Christensenella.

The goal of this observational study is to constitute a biological samples collection from centenarian people, to proceed with the isolation of beneficial commensal strains such as Faecalibacterium prausnitzii, Akkermansia muciniphila and Oscillospiraceae, in a non-limitative way.

Elderly and centenarian people will be recruited in nursing home among the Gerontopole of "Ile de France" network.

Blood (serum + TruCulture tubes) and stools will be collected from each subject.

ELIGIBILITY:
Inclusion Criteria:

* 95 years and older
* BMI between 18.5 and 25 kg/m2
* Clinical exam normal
* Subject agreeing to participate in the study and not objecting to participate in the study.
* Able and willing to provide samples of blood and faeces

Exclusion Criteria:

* Diagnosed acute or chronic gastrointestinal disease or complication (e.g., celiac disease, gastroesophageal reflux, gastric or duodenal ulcer, Crohn's disease, hemorrhoids, irritable bowel syndrome)
* Infectious gastrointestinal event within 3 months prior to inclusion
* Diabetes
* Severe chronic disease (active cancer, HIV, severe renal failure, ongoing severe heart or liver or biliary disorders, arthritis) or severe chronic disease deemed incompatible with the conduct of the study by the investigator
* Major surgical procedure likely to disrupt the intestinal microbiota, within 6 months prior to inclusion
* Recent food allergy < 3 months prior to inclusion
* Antibiotic, antiviral, antifungal, proton pump inhibitor or any other treatment likely to disrupt the microbiota in the 3 months prior to inclusion
* Previous or current use of a treatment that may disrupt the microbiota (e.g. laxatives, antidiarrheals, antacids...) in the last 3 months
* Significant change in dietary habits or physical activities in the 3 months prior to inclusion
* Consumption of more than 2 standard glasses of alcoholic beverages per day
* Smoking > 20 cigarettes per day, illicit drug use,
* Daily use of non-steroidal anti-inflammatory drugs (NSAIDs)
* Severe psychiatric or neurological pathology
* Completely dependent subject (GIR Score = 1)
* Subject with liquid stools (Bristol Score = 7) or very hard stools (Bristol Score = 1)
* Vaccination in the last month before inclusion
* Subject unable to understand the purpose of the research, answer questions and give their decision to participate in the study
* Subject already included in another research study involving the human subject
* Subject under guardianship and whose guardianship objects to the participation of his/her protectee,
* Subject not affiliated with a social security plan or not a beneficiary of such a plan

Min Age: 95 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Study Population: Elderly (>95 years old) and centenarians people
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Establishment of a bank of blood and faeces biological samples from centenarians people for research purposes | One day
  Study will collect up to 18 mL of blood and minimum of 20g of faeces at one visit from people aged > 95 years.

SECONDARY OUTCOMES:
Bacteria collection | One day
  Isolation and culture of bacteria of interest
Fecal microbiota composition | One day
  Measures of alpha and beta diversity of fecal samples
Immuno-modulatory properties of isolated strains | One day
  Cellular assays with immune related readout to decipher pro and/or anti inflammatory properties

CONTACTS AND LOCATIONS:
Overall Officials: Cyril GUYARD, Study Director — Bioaster; Olivier HANON, Principal Investigator — Gérond'if
Locations (1):
- Gerond'if - Gérontopôle Ile de France, Paris, France

IPD SHARING:
Plan to Share IPD: No